CLINICAL TRIAL: NCT00804154
Title: A Phase I Study of the Intrathecal Administration of Resiniferatoxin for Treating Severe Refractory Pain Associated With Advanced Cancer
Brief Title: Resiniferatoxin to Treat Severe Pain Associated With Advanced Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090039; 09-N-0039
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-12-16

CONDITIONS: Intractable Pain; Palliative Care
Keywords: Vanilloid; Capsaicin; Cancer Pain; Nerve Block
MeSH Terms: conditions — Pain, Intractable; Cancer Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): advanced cancer patients with pain
  Interventions: Drug: Intrathecal Resiniferatoxin

INTERVENTIONS:
Drug: Intrathecal Resiniferatoxin — phase I, single-site, non-randomized, open-label, dose-escalation study to determine the safety and efficacy of IT RTX in subjects with severe refractory pain due to advanced malignancy

SUMMARY:
This study will examine the safety of giving the experimental drug, resiniferatoxin (RTX), to treat severe pain in patients with advanced cancer. RTX is a chemical extracted from a cactus-like plant. It is similar to capsaicin, the active ingredient in hot pepper. RTX has relieved pain and reduced the need for pain medication in several animal experiments. It works by destroying nerves that transmit pain information.

People at least 18 years of age with severe pain from advanced cancer at or below the level of the chest that cannot be controlled with standard treatments may be eligible for this study. Participants undergo the following procedures:

Pretreatment Visit

Before beginning treatment with RTX, patients give a medical history and undergo a physical examination that includes:

* Electrocardiogram (EKG)
* Blood draw
* Urinalysis
* Neurological examinations
* Peak expiratory flow rate (PEFR)
* Eye examination
* MRI
* Urology assessment
* Pregnancy test, when appropriate
* Questionnaires to collect information on health, personality, mood, pain levels and symptoms.

  2-Day Hospitalization

Patients are hospitalized for 2 days for RTX injection and monitoring, as follows:

* RTX injection: RTX is injected in the operating room under general anesthesia. It is given through a catheter placed in the patient s spine. The catheter is also used to obtain samples of cerebrospinal fluid (CSF) the clear fluid that bathes the spinal cord. The fluid is examined to assess drug effects and side effects, chemical changes in the content of the CSF associated with RTX, and how RTX is handled by the body.
* Post-injection monitoring, including:
* Surveys about symptoms such as pain or weakness
* Neurological examinations
* Blood and CSF sampling
* EKG
* AEs

Outpatient followup

* Vitals
* Blood draw, Urinalysis, neurological and sensory testing, EKG on days 7, 14 and 30 after the injection
* MRI scans of the head and back, Urology assessment and PEFR on day 15 after the injection
* Eye examination
* Follow-up phone calls monthly for 6 months

DETAILED DESCRIPTION:
Pain continues to be a major problem in patients with advanced cancer. Resiniferatoxin (RTX), a potent member of the family of drugs that includes capsaicin, selectively and irreversibly destroys the neurons (or their axons) transmitting chronic pain sensation. Intrathecal injection of RTX in several animal species has demonstrated a high level of safety, specificity, and efficacy in treating severe pain. This first-in-human, dose-escalation study is investigating the intrathecal administration of RTX in cancer patients with severe pain.

PRIMARY OBJECTIVE:

To investigate the safety and efficacy of RTX administered intrathecally in subjects with severe refractory pain associated with advanced cancer.

STUDY POPULATION:

Up to 45 subjects will be accrued. Eligible subjects will be greater than or equal to 18 years of age, have a clinical and histological diagnosis of advanced malignancy, and have severe pain due to malignancy that is at or below the level of the chest and not adequately relieved by other pain control therapies.

DESIGN:

This is a single site, non-randomized, open-label, dose-escalation study using a modified Fibonacci scheme. The starting dose of RTX was 13 micrograms given as a 2 mL injection via an intra-spinal catheter over approximately 30 seconds followed by a 1 mL flush. Six subjects were dosed at this level and 3 were dosed at the 26 microgram dose level at the same volume of injectate, flush and injection time. Under the study design, RTX doses were to be increased in progressively smaller percentage increments with each dose-escalation to occur in sequential groups of 3 subjects until 1 escalation above the effective dose in 100% of subjects (ED100), completion of the 100 microgram dose level, or establishment of the maximum tolerated dose (MTD), whichever occurs first. The total duration of study participation for any subject will be up to 7 months.

The amended RTX injection technique reduced the injection volume and increased the injection time to reduce the spread of RTX to above the T6 (sixth thoracic) vertebral level. The present technique is a 1 mL injection over 2 minutes (0.5 mL/minute) given via infusion pump, followed by flushing of the IT catheter with the minimum volume of sterile, preservative-free saline necessary to clear the internal volume of the catheter used for the injection. Three patients were treated at the new starting dose of 13 micrograms with the new injection technique. The next 3-patient cohort will receive a dose of 26 micrograms. The subsequent subject dose tier will receive a dose of 44 micrograms consistent with the protocol s dose-escalation algorithm. Administering this dose will require an infusion volume of 1.76 mL of the present 25 micrograms/mL RTX formulation.

OUTCOME MEASURES:

The primary study outcome is the ED100, the MTD, or the maximum dose administered, whichever is achieved first during dose-escalation. The primary pain variable for determining the ED100 is the daily worst pain intensity score averaged over a 4 to 7-day period during the 3 weeks before RTX dosing and during Days 8 through 14 after dosing. The numerical rating scale (NRS), administered verbally during a daily telephone interview, will be the primary pain assessment instrument. For a given subject, the treatment will be considered effective if the subject experiences a greater than or equal to 50% reduction in the mean daily worst pain score assessed by NRS (evaluated on Study Day 15). We may also consider RTX treatment to be successful if there is greater than or equal to 50% reduction in opiate intake, measured by morphine milligram equivalents (MME) per day, even if pain levels are unchanged after RTX treatment.

Secondary outcome measures will be other surveys of pain, including an assessment of worst daily pain by the visual analog scale, and assessments of function and quality of life.

Safety assessments will include hematology; serum clinical chemistry tests; cerebrospinal fluid examinations; physical, neurological, and eye examinations; reporting of adverse events; electrocardiograms; and findings on magnetic resonance imaging of the spine and brain.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subject inclusion criteria are based on inadequate control of pain despite best efforts, including appropriate use of analgesic medications. To be enrolled in the study, subjects must meet all of the following criteria:

1. Age 18 years or older.
2. Clinical and histological diagnosis of cancer with disease that has not adequately responded to standard therapies. A pathology report documenting malignancy is required.
3. Subject not currently seeking or receiving potentially curative therapies for cancer (e.g., chemotherapy or immunotherapy). Curative cancer therapy may be sought after the Day 15 clinic visit, and palliative anti-tumor therapy is allowed as long as the subject was established on that therapy prior to enrollment (see exclusion criterion 6).
4. Mean daily worst pain NRS score of greater than or equal to 6 for pain at or below the T6 dermatome (level of the chest) that is associated with a malignant disease. The mean score must be derived from recordings on at least 4 of 7 consecutive days within 3 weeks preceding treatment.
5. Alternative methods of pain control are not sufficiently effective, not indicated, not tolerated, and/or refused by the subject, as determined by the Pain and Palliative Care Service (PPCS). Alternative methods of pain control include, but are not limited to, the following:

   -Opioids (all routes of administration including neuraxial infusions)

   -Adjuvant pain medications such as antidepressants, corticosteroids, local anesthetics, and antiseizure medications

   -Procedures such as catheter or implantable pump placement for delivery of analgesic medication
   * Prior neurolytic interventions (including intercostal, superior hypogastric, or celiac plexus blocks)
   * Complementary medicine approaches
   * Transcutaneous electric nerve stimulation
   * Radiation therapy
6. Reasonable expectation that the subject will be able to complete the study through the 30-day follow-up.
7. Medical clearance from referring physician consisting of a statement indicating an adequate recovery period from other previous trials/medication.
8. Formal review of the subject s medical records and written approval for his/her inclusion in

the study by 3 separate persons:

* Principal Investigator (PI) or an Associate Investigator (AI)
* Medical oncologist or oncologic surgeon.
* A member of the PPCS at the NIH or institution s equivalent at other sites.

  10. International normalized ratio (INR; from prothrombin time [PT]) < 1.5 and partial thromboplastin time (PTT) less than or equal to the upper limit of the reference range. The INR and PTT may be corrected (e.g., by administration of blood products, vitamin K, etc.), provided a repeat blood draw confirms that the values meet this inclusion criterion.

  10. Platelet count greater than or equal to 50,000/mm^3. Platelets will be transfused as necessary to raise the platelet count to greater than or equal to 100,000/mm^3 prior to dosing.

  11. Ability to stop any anticoagulant (e.g., Coumadin) and antiplatelet therapies (e.g., aspirin) before and during IT catheter placement according to accepted medical guidelines.1

  12. Ability and willingness to undergo an eye examination.

  13. Ability to read, speak, and understand English, and willingness to complete the study tools and forms.

  14. For women of childbearing potential and men with partners of childbearing potential, the ability and willingness to use an effective method of contraception during the study. Effective methods of birth control include:
* hormonal contraception (birth control pills, injected hormones, or vaginal ring),
* intrauterine device,
* barrier methods (condom or diaphragm) combined with spermicide, or
* surgical sterilization (hysterectomy, tubal ligation, or vasectomy).

  15. Availability of a responsible adult to assist with activities of daily living as needed for the subject through the Day 15 visit.

  16. Ability to assign a Durable Power of Attorney (DPA) for research and medical care at NIH

EXCLUSION CRITERIA:

Subjects will be excluded from the study if they meet any of the following criteria:

1. Primary pain source from anatomical regions at T5 dermatome or above.
2. Pain due to causes other than cancer or its treatment that is moderate to severe in intensity.
3. Anatomic abnormality or pathology of the spinal cord and/or IT space on magnetic resonance imaging (MRI) that could increase the risk of adverse effects of catheter placement or interfere with CSF flow.
4. Evidence of advanced brain pathology or elevated intracranial pressure as determined by symptoms, history, physical examination (including neurological and eye examination), and/or MRI.
5. Presence of an IT shunt device (e.g., ventriculo-peritoneal and ventriculo-atrial shunts).
6. Anticipating initiation of palliative anti-tumor therapy or significant changes to current palliative anti-tumor therapy before completion of the Day 15 visit.
7. Documented allergy to chili peppers or capsaicin (e.g., hives, wheal).
8. Contraindication to MRI or MRI contrast.
9. Female subjects who are pregnant or lactating.
10. Clinically significant disorder or condition that might interfere with study participation or greatly increase safety risk to the subject, as judged by a study investigator.
11. Planned use of another investigational agent, therapy, or device within 30 days after dosing.
12. Have a history of heart failure or unexplained fainting (syncope).
13. Have an EKG abnormality in which the baseline QTc interval exceeds 450 milliseconds.
14. Have a known family history of long QT syndrome.
15. Have abnormal electrolyte levels (i.e., low potassium) that cannot be corrected.
16. Have urinary retention that does not resolve with medical or surgical treatment.
17. Have skin ulceration that does not resolve with medical or surgical treatment.
18. Have a history of seizure activity in the previous month.
19. Have experienced symptoms of opioid toxicity in the past month (i.e. myoclonus, seizures, and/or hallucinations)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2009-08-14 (Actual); Primary Completion 2026-02-07 (Estimated); Study Completion 2026-02-07 (Estimated)

PRIMARY OUTCOMES:
Investigate the safety and efficacy of RTX administered intrathecally in subjects with severe refractory pain associated with advanced cancer along with ED100, the MTD, or the maximum dose administered, whichever is achieved first during dose es... | Day 7, Day 15, Day 68, Day 188
  Dose escalation decisions are based on both effectiveness (as assessed by mean worst pain on the NRS) and DLT. The dose escalation population will include all subjects who are dosed, complete the NRS, and have the DLT assessments from baseline through Day 15. Subjects who are not evaluable for dose escalation will be replaced.

SECONDARY OUTCOMES:
Secondary outcome measures will be other surveys of pain, including an assessment of worst daily pain by the visual analog scale, and assessments of function and quality of life. | Day 7, Day 15, Day 68, Day 188
  The secondary outcome variables will be summarized over time by dose cohort as appropriate for the outcome measure. Absolute and percentage change in the NRS and VAS pain scores between the pre- and post-RTX dosing assessments (baseline period and study Days 8 through 14, respectively) will also be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: John D Heiss, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do plan to share IPD. we will share all IPD that results in a publication on a public repository, as required by most journals. the data will be de-identified and anonymized.

REFERENCES:
- [Background] Daut RL, Cleeland CS. The prevalence and severity of pain in cancer. Cancer. 1982 Nov 1;50(9):1913-8. doi: 10.1002/1097-0142(19821101)50:93.0.co;2-r. PMID 7116316
- [Background] Cleeland CS, Gonin R, Hatfield AK, Edmonson JH, Blum RH, Stewart JA, Pandya KJ. Pain and its treatment in outpatients with metastatic cancer. N Engl J Med. 1994 Mar 3;330(9):592-6. doi: 10.1056/NEJM199403033300902. PMID 7508092
- [Background] Oster MW, Vizel M, Turgeon LR. Pain of terminal cancer patients. Arch Intern Med. 1978 Dec;138(12):1801-2. PMID 718345
- [Derived] Mannes AJ, Heiss JD, Berger A, Alewine CC, Butman JA, Hughes MS, Rabbee N, Hayes C, Williams TS, Sapio MR, Iadarola MJ. Treatment of Intractable Cancer Pain with Resiniferatoxin - An Interim Study. NEJM Evid. 2025 Jun;4(6):EVIDoa2400423. doi: 10.1056/EVIDoa2400423. Epub 2025 May 27. PMID 40423401
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2009-N-0039.html